CLINICAL TRIAL: NCT00908011
Title: A Prospective, Randomized Study to Determine the Effect of Ezetimibe in Addition to Rosuvastatin on Lipids in Participants With the Hypercholesterolemia Associated With HIV Antiretroviral Therapy
Brief Title: Addition of Ezetimibe (Ezetrol®) to Ongoing Therapy With Rosuvastatin (Crestor®) in HIV Positive Patients Not Reaching Cholesterol Targets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Merck Frosst-Schering Pharma, G.P. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H08-00287
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-11

CONDITIONS: Hypercholesterolemia; HIV Infections
Keywords: Hypercholesterolemia; HIV; Ezetimibe; Statin; Apolipoprotein B100/Apolipoprotein A1 ratio
MeSH Terms: conditions — Hypercholesterolemia; HIV Infections | interventions — Ezetimibe; Rosuvastatin Calcium; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe (Active Comparator): 10mg/day ezetimibe in addition to ongoing rosuvastatin treatment (10mg/day)
  Interventions: Drug: Ezetimibe
- Standard Care (Active Comparator): Increased dose of rosuvastatin to 20mg/day
  Interventions: Drug: Rosuvastatin (standard care)

INTERVENTIONS:
Drug: Ezetimibe — 10mg/day ezetimibe in addition to ongoing rosuvastatin treatment (10mg/day)- tablet, orally, 10mg/day for 12 weeks
  Other Names: Ezetrol
  Arms: Ezetimibe
Drug: Rosuvastatin (standard care) — Increased dose of rosuvastatin to 20mg/day
  Other Names: Crestor
  Arms: Standard Care

SUMMARY:
This study involves comparing the effectiveness of treatments in HIV positive patients who may be predisposed to heart attack or stroke. The investigators will evaluate the effectiveness of two drugs, often prescribed by doctors to these patients, at lowering cholesterol and thereby making the patient less them less vulnerable to suffering a heart attack or stroke. The investigators believe that the addition of a second drug, from a different class of cholesterol lowering medications, will improve the outcome of the patients by lowering cholesterol.

DETAILED DESCRIPTION:
This study seeks to determine whether HIV positive patients who have suboptimal lipids and/or are not reaching specified lipid targets will benefit from the addition of a second lipid lowering drug (ezetimibe) to existing lipid lowering therapy with a statin (specifically rosuvastatin) versus increasing the dose of the ongoing statin in terms of improvements in serum lipid parameters namely total cholesterol, LDL, HDL, triglycerides and apolipoprotein B100 (apoB), apolipoprotein A1 (apoA1), apoB/apoA1 ratio.

The target population will be HIV+ patients with hypercholesterolemia due to highly active antiretroviral therapy, the study will have a randomized, parallel design. Sample size will be 50 patients already taking 10 mg of rosuvastatin who are not reaching lipid targets to receive either an increased dose of rosuvastatin (20mg) or to receive 10mg ezetimibe in addition to their ongoing rosuvastatin therapy. There will be 25 patients randomized to each group.

At baseline serum samples will be obtained and tested for serum triglycerides, total cholesterol, HDL, total cholesterol:HDL ratio, apoB, apoA1, apoB/apoA1 ratio, liver transaminases (AST and ALT), CK, thyroid stimulating hormone, creatinine and fasting blood glucose.

After 12 weeks of therapy serum samples will once again be obtained and tested for serum triglycerides, total cholesterol, HDL, total cholesterol:HDL ratio, apolipoprotein B100, liver transaminases (AST and ALT), CK, thyroid stimulating hormone, creatinine and fasting blood glucose.

The primary hypothesis is that the combination of rosuvastatin and ezetimibe will lower serum apolipoprotein B100/apolipoprotein A1 ratio more so than an increased dose of rosuvastatin alone, in participants with mixed dyslipidemia associated with HIV therapy.

Secondarily we believe the combination of rosuvastatin and ezetimibe will lower the concentrations of serum cholesterol, LDL-cholesterol, triglycerides, apolipoprotein B100 and C-reactive protein more so than an increased dose of rosuvastatin alone, and that there will be no increase in side effects when administered to participants with mixed dyslipidemia associated with HIV therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* currently taking 10mg of rosuvastatin
* recent (within three months) fasting lipid profile in which the serum total cholesterol to HDL ratio is >5.0

Exclusion Criteria:

* Previous adverse reaction to ezetimibe
* taken ezetimibe within 30 days of starting the study
* history of vascular disease
* allergic reaction or muscle problems while taking any statin
* currently taking other lipid lowering medications (i.e. a fibrates or cholestyramine)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-06; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Bondy, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital HIV Immunodeficiency/Metabolic Clinic, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ezetimibe | Standard Care
Started | 23 | 20
Completed | 21 | 18
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe | Standard Care | Total
Number analyzed (Participants) | 23 | 20 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 20 | 43
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (7.4) | 57.0 (9.9) | 57 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 22 | 17 | 39
Region of Enrollment [Number; unit: participants]
  Canada | 23 | 20 | 43

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Difference in Final Value of Serum Apolipoprotein B Between Participants Treated With Rosuvastatin Versus Participants Treated With Both Rosuvastatin and Ezetimibe.
Time Frame: 3 months from baseline
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ezetimibe | Standard Care
Number analyzed (Participants) | 21 | 18
mmol/L | 0.88 (0.22) | 0.89 (0.25)

2. Secondary Outcome: Percent Change in Apolipoprotein B, Percent and Absolute Change Total Cholesterol, LDL, HDL, Triglycerides, Apolipoprotein A1, apolipoproteinB/apoliporoteinA1 Ratio and C-reactive Protein
Time Frame: 3 months from baseline
Reporting Status: Not Posted

3. Secondary Outcome: Assessment of Safety Parameters, Specifically Incidence of Complications as Measured by an Increase in AST &/or ALT ≥3-fold ULN & a CK ≥10-fold ULN
Time Frame: 3 months from baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ezetimibe | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No